CLINICAL TRIAL: NCT02269202
Title: Pharmacokinetics of 7.5 mg Midazolam, Given Orally With and Without Concomitant Administration of 175 mg Crobenetine, Given as a 6 Hrs i.v. Infusion (One Hour Loading Dose Directly Followed by a Five Hours Maintenance Dose). A Randomised, Single Blind, Two-way Crossover Trial in Healthy Male Subjects
Brief Title: Pharmacokinetics of Midazolam, With and Without Concomitant Administration of Crobenetine in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Single | Purpose: Treatment
Other Study IDs: 599.12
Record Dates: First submitted 2014-10-16; First posted 2014-10-21 (Estimated); Last update posted 2014-10-21 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
MeSH Terms: interventions — Midazolam; BIII 890 CL

ARMS (2):
- Midazolam and crobenetine (Experimental)
  Interventions: Drug: Midazolam, tablet; Drug: Crobenetine, i.v. infusion
- Midazolam and placebo (Placebo Comparator)
  Interventions: Drug: Midazolam, tablet; Drug: Placebo

INTERVENTIONS:
Drug: Midazolam, tablet
Drug: Crobenetine, i.v. infusion
  Arms: Midazolam and crobenetine
Drug: Placebo
  Arms: Midazolam and placebo

SUMMARY:
To assess the pharmacokinetics of midazolam with/without concomitant administration of crobenetine

ELIGIBILITY:
Inclusion Criteria:

- All participants in the study should be healthy males, range from 21 to 50 years of age and their bodymass index (BMI) be within 18.5 to 29.9 kg/m2

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy), which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (> 24 hours) within at least one month or less than ten half-lives of the respective drug before enrolment in the study (except substitution therapy regarding thyroid gland)
* Use of any drugs that might influence the results of the trial (within one week prior to administration or during the trial)
* Participation in another trial with an investigational drug (within two months prior to administration or during the trial)
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Blood donation (≥ 100 mL, within four weeks prior to administration or during the trial)
* Excessive physical activities (within the last week before the study)
* Any laboratory value outside the reference range of clinical relevance

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2002-02; Primary Completion 2002-04 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of midazolam from zero time extrapolated to infinity (AUC0-infinity) | up to 24 hours after start of drug administration
Maximum observed concentration of midazolam in plasma (Cmax) | up to 24 hours after start of drug administration

SECONDARY OUTCOMES:
Area under the concentration-time curve (AUC) | up to 24 hours after start of drug administration
Time to maximum observed concentration (tmax) | up to 24 hours after start of drug administration
Individual time courses of plasma concentrations | up to 24 hours after start of drug administration
Terminal rate constant in plasma (λz) | up to 24 hours after start of drug administration
Terminal half-life in plasma (t1/2) | up to 24 hours after start of drug administration
Mean residence time in the body (MRT) | up to 24 hours after start of drug administration
Apparent clearance in plasma (CL/F) | up to 24 hours after start of drug administration
Volume of distribution (V) | up to 24 hours after start of drug administration
Changes from baseline in physical examination | pre-dose and day 8 after drug administration
Number of patients with clinically relevant findings in vital signs | up to day 8 after drug administration
  blood pressure, pulse rate
Number of patients with clinically relevant findings in 12-lead ECG | up to day 8 after drug administration
Number of patients with clinically relevant findings in laboratory tests | up to day 8 after drug administration
Number of patients with adverse events | up to day 8 after drug administration
Global assessment of tolerability by the investigator on a 4-point rating scale | up to 192 hours after start of drug administration